CLINICAL TRIAL: NCT04818918
Title: Study of the Relationship Between Coronary Flow and Myocardial Viability: the Single-centre, Observational, Prospective FloVITA Study
Brief Title: Coronary Flow and Myocardial Viability: the FloVITA Study
Acronym: FloVita
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0123456
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Myocardial Infarction; Myocardial Ischemia
Keywords: microvascular resistance; fractional flow reserve; myocardial viability
MeSH Terms: conditions — Myocardial Infarction; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STEMI group: Patients with anterior ST segment MI treated with percutaneous coronary intervention of the left anterior descending artery, at least 7 days prior to inclusion, and scheduled for new angiography to evaluate FFR of a lesion other than the infarct-related artery.
  Absolute coronary flow and microvascular resistance will be measured in the LAD.
  Interventions: Device: Absolute coronary flow measurement; Device: Microvascular resistance measurement; Other: Cardiac MRI
- Control group: Patients undergoing non-urgent coronary angiography for stable angina or silent ischemia, with measure of FFR on one or more vessels (intermediate lesions <90% without proven ischemia). Absence of any signfiicant lesion on the left anterior descending artery (as evaluated by angiography or FFR value >0.8).
  Absolute coronary flow and microvascular resistance will be measured in the LAD.
  Interventions: Device: Absolute coronary flow measurement; Device: Microvascular resistance measurement

INTERVENTIONS:
Device: Absolute coronary flow measurement — Absolute coronary flow will be measured.
Device: Microvascular resistance measurement — Microvascular resistance will be measured.
Other: Cardiac MRI — Cardiac MRI will be performed to evaluate myocardial viability.
  Groups: STEMI group

SUMMARY:
Evaluation of fractional flow reserve (FFR) is a key method for assessing ischemia with a view to guiding revascularization strategy following acute coronary syndrome. A stenosis that appears to be severe by angiography may cause limited ischemia (with an FFR value >0.80) due to the incapacity of the necrotic zone to achieve physiological hyperemia, i.e. maximal coronary flow. Recently, it has been demonstrated that absolute coronary flow, and micro- and macrovascular resistance, as measured by a thermodilution technique, using the Rayflow microcatheter (Hexacath) are strongly associated with myocardial mass. In extensive necrosis, there is a loss of myocardial mass, and these tools could be of potential interest in measuring myocardial viability, which reflects the extent of remaining viable myocardial mass.

Therefore, this study aims to investigate the relationship between both absolute coronary flow and microvascular resistance, and myocardial viability assessed by MRI.

In a prospective, single-centre, interventional study, we will compare absolute coronary flow and microvascular resistance in the left anterior descending artery, in patients with and without a history of ST segment elevation MI.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the STEMI group:

  * ST segment elevation MI ≥7 days treated by angioplasty of the left anterior descending (LAD) artery
  * Scheduled to undergo angiography for fractional flow reserve (FFR) assessment of a lesion other than the infarct-related artery.
* Inclusion criteria for the control group:

  * patients undergoing non-urgent coronary angiography for stable angina or silent ischemia
  * with measure of the FFR on one or more vessels (intermediate lesion <90% without proven ischemia)
* absence of any significant lesion on the LAD (as assessed by angiography or FFR>0.8)
* Inclusion criteria for both groups:

  * Written informed consent
  * Affiliation to a social security regimen (or beneficiary thereof).

Exclusion Criteria:

* Target vessel (LAD) not permeable.
* FFR <0.8 in the LAD
* Coronary spasm
* Left ventricular ejection fraction <0.50 or a history of anterior MI in patients in the control group
* Hypertrophic cardiomyopathy
* Severe valvular heart disease
* History of coronary artery bypass graft
* Patients with limited legal capacity or patients under guardianship/tutorship
* Patients with anticipated poor compliance as assessed by the investigator
* Patients not affiliated to any social security regime.
* Pregnant women.
* Subjects within the exclusion period of another clinical trial as noted in the national registry of research volunteers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recent (>=7 days) ST segment elevation MI for the intervention group, and patients with stable angina or silent ischemia for the control group.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2021-05-19 (Actual); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Coronary flow (mL/min) in the LAD | At the end of the angiography procedure
  Measurement of coronary flow in mL/min in the left anterior descending artery

SECONDARY OUTCOMES:
Microvascular resistance | At the end of the angiography procedure
  Measurement of microvascular resistance in the LAD
Myocardial necrosis | Cardiac MRI to be performed 7 to 30 days after index angiography procedure
  Extent of myocardial necrosis on cardiac MRI (number of segments)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Meneveau, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- CHU Besancon, Besançon, France

REFERENCES:
- [Derived] Guillon B, Besutti M, Revel L, Seronde MF, Meneveau N, Chopard R. Absolute Coronary Flow Reduction Mediated by Microvascular Resistance in Myocardial Infarction: The FLOVITA Study. Catheter Cardiovasc Interv. 2025 Dec;106(7):3588-3596. doi: 10.1002/ccd.70268. Epub 2025 Oct 13. PMID 41078218